CLINICAL TRIAL: NCT03906110
Title: Community Colorectal Cancer Awareness, Research, Education & Screening (C-CARES) : A Multilevel Intervention to Increase Colorectal Cancer Screening Adherence In Community Clinics
Brief Title: Community Colorectal Cancer Awareness, Research, Education & Screening (C-CARES)
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: MCC-19106
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer Screening; FIT test; Fecal Immunochemical Test
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Educational Status; Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- C-Cares: Participants will be given Community Colorectal Cancer Awareness, Research, Education and Screening (C-CARES) Materials and FIT kits.
  Interventions: Behavioral: Community Colorectal Cancer Awareness, Research, Education & Screening (C-CARES) Materials; Behavioral: Contact Message; Diagnostic Test: Fecal Immunochemical Test (FIT)
- C-Cares Plus: Participants will be given Community Colorectal Cancer Awareness, Research, Education and Screening (C-CARES) materials, FIT kits, and personalized one-on-one education and coaching.
  Interventions: Behavioral: Community Colorectal Cancer Awareness, Research, Education & Screening (C-CARES) Materials; Behavioral: Contact Message; Behavioral: Personalized One on One Education; Diagnostic Test: Fecal Immunochemical Test (FIT)

INTERVENTIONS:
Behavioral: Community Colorectal Cancer Awareness, Research, Education & Screening (C-CARES) Materials — Educational materials (photonovella +DVD) + Fecal Immunochemical Test (FIT) kit. Offers colorectal cancer screening information using a novella format. Materials describe colorectal cancer and screening tests that are available, and procedures for completing FIT kit.
Behavioral: Contact Message — Card with a general message about colorectal cancer screening. This same message will be delivered at 3 time points.
Behavioral: Personalized One on One Education — * Trained study coordinators will meet with participant for a brief 15 minute educational session delivered in clinic that summarizes information from the materials and demonstrates FIT collection.
  * Email or text reminders with brief messages in clear language will be sent that aim to remind and prompt patients to complete FIT.
  * For participants that are not responsive to above, trained study staff will address specific FIT specific hinderances by telephone or in clinic.
  * Participants will receive a one page summary of key points of salience of repeat screening "GET FIT AGAIN". Another FIT kit is provided.
  Groups: C-Cares Plus
Diagnostic Test: Fecal Immunochemical Test (FIT) — The Fecal Immunochemical Test (FIT), is a screening test that detects hemoglobin in stool samples, only requiring one stool sample.

SUMMARY:
The purpose of this study is to test if including personalization in education materials about colorectal cancer screening is more effective at helping encourage people to complete colorectal cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand, read and speak English or Spanish
* Are not up-to-date with colorectal cancer screening
* No symptoms of colorectal cancer
* Not at increased risk for colorectal cancer due to family history or personal high-risk GI syndromes

Exclusion Criteria:

* Symptoms of colorectal cancer
* Family history of colorectal cancer

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Established patients of community health clinics aged 50-75 with average risk of colorectal cancer.
Sampling Method: Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Fecal Immunochemical Test (FIT) use -Time Point 1 | Time Point 1 (at 3 months)
  Participants use of FIT kits will be measured based on FIT sample return rate.
Fecal Immunochemical Test (FIT) Use- Time Point 2 | Time Point 2 (up to 18 months)
  Participants use of FIT kits will be measured based on FIT sample return rate.
Fecal Immunochemical Test (FIT) Use- Time Point 3 | Time Point 3 (End of study, up to 30 months)
  Participants long term FIT adherence will be measured based on FIT sample return rate.

CONTACTS AND LOCATIONS:
Overall Officials: Clement K Gwede, PhD, MPH, RN, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christy SM, Sutton SK, Abdulla R, Boxtha C, Gonzalez P, Cousin L, Ewing A, Montoya S, Lopez D, Beehler T, Sanchez J, Carvajal R, Meade CD, Gwede CK. A multilevel, low literacy dual language intervention to promote colorectal cancer screening in community clinics in Florida: A randomized controlled trial. Prev Med. 2022 May;158:107021. doi: 10.1016/j.ypmed.2022.107021. Epub 2022 Mar 17. PMID 35305995